CLINICAL TRIAL: NCT04063670
Title: Coping After Pediatric Scoliosis Surgery: How Does it Affect Pain and Function?
Brief Title: Coping After Pediatric Scoliosis Surgery
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-26617
Record Dates: First submitted 2019-05-11; First posted 2019-08-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Pain; Function; Pediatric; Scoliosis; Scoliosis Surgery; Spinal Fusion; Idiopathic Scoliosis; Coping; Coping Skills; Education; Video Intervention; Randomized; Prospective; Satisfaction; Adolescent; Opioid
MeSH Terms: conditions — Pain; Scoliosis; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized Controlled Clinical Trial
Who Masked: Care Provider
Masking Description: All clinicians and care providers are blinded to participants randomized group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Routine, standard-of-care treatment
  Interventions: Other: Control
- Video Intervention (Experimental): Routine, standard-of-care PLUS peri-operative video series
  Interventions: Other: Video Intervention

INTERVENTIONS:
Other: Video Intervention — Peri-operative video series focusing on expanded education and coping skills before and after scoliosis surgery for adolescent idiopathic scoliosis
  Arms: Video Intervention
Other: Control — Routine, Standard-of-Care
  Arms: Control

SUMMARY:
This is a prospective, randomized controlled trial evaluating the efficacy of expanded patient education and coping skills on pain management following multilevel pediatric spinal surgery. The intervention will include a smartphone- based platform and a comprehensive library of peri-operative educational and coping skills videos as a means for better addressing the psychosocial elements of a child's individual pain experience. The study evaluated whether this novel intervention will reduce pain, improve outcomes and accelerate functional recovery up to 6 weeks after surgery.

ELIGIBILITY:
Inclusion criteria:

- All children ages 11 to 18 years old treated with primary multilevel spinal surgery of any approach

Exclusion Criteria:

* Non-English speaking
* Non-idiopathic scoliosis, such as neuromuscular, congenital or syndromic.
* Other comorbidity, including developmental delay.
* Any surgical complication that results in significant divergence from our institution's standard scoliosis pathway.
* Unplanned admission within 6 weeks of index operation.
* Active treatment psychotherapy and/or cognitive behavioral therapy for any reason

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Post-Operative Pain | Up to 6-weeks post-operatively
  Outcome #1 will evaluate the intervention's impact on post-operative pain via completion of the computer-adaptive NIH PROMIS measures on pain intensity and pain behavior.
  For each of the PROMIS measures, a score of 50 is the average for the United States general population with a standard deviation of 10. All scores are converted to T-scores. The T-score and standard error are automatically reported after completion of the computer-adaptive test. A higher PROMIS T-score represents more of the concept being measured. As each patient will have a pre-operative baseline score, the difference between pre- and post-operative scores will be utilized for all further analysis, with a difference of 10 points (1-standard deviation) scored as the minimal clinically significant difference.
Post-Operative Pain | Up to 6-weeks post-operatively
  Outcome #2 will evaluate the intervention's impact on a proxy for post-operative pain via completion of a 1-question survey on recent opioid consumption. The question is formatted as a 5-point Likert scale, scored 1-5, with higher scores indicating more frequent opioid consumption.

SECONDARY OUTCOMES:
Patient Reported Outcomes - Global Health | Up to 6-weeks post-operatively
  Outcome #3 will measure patient reported outcomes via administration of the computer adaptive NIH PROMIS measures for global health.
  For each of the PROMIS measures, a score of 50 is the average for the United States general population with a standard deviation of 10. All scores for this measure will be converted to T-scores via the NIH's published guidelines. As each patient will have a pre-operative baseline score, the difference between pre- and post-operative scores will be utilized for all further analysis, with a difference of 10 points (1-standard deviation) scored as the minimal clinically significant difference.
Patient Reported Outcomes - Mobility | Up to 6-weeks post-operatively
  Outcome #4 will measure patient reported outcomes and functional status via completion of the computer-adaptive NIH PROMIS measure for mobility
  For each of the PROMIS measures, a score of 50 is the average for the United States general population with a standard deviation of 10. All scores are converted to T-scores. The T-score and standard error are automatically reported after completion of the computer-adaptive test. A higher PROMIS T-score represents more of the concept being measured. As each patient will have a pre-operative baseline score, the difference between pre- and post-operative scores will be utilized for all further analysis, with a difference of 10 points (1-standard deviation) scored as the minimal clinically significant difference.
Patient Reported Outcomes - Positive Affect | Up to 6-weeks post-operatively
  Outcome #5 will measure patient reported outcomes via completion of the computer-adaptive NIH PROMIS measure for positive affect.
  For each of the PROMIS measures, a score of 50 is the average for the United States general population with a standard deviation of 10. All scores are converted to T-scores. The T-score and standard error are automatically reported after completion of the computer-adaptive test. A higher PROMIS T-score represents more of the concept being measured. As each patient will have a pre-operative baseline score, the difference between pre- and post-operative scores will be utilized for all further analysis, with a difference of 10 points (1-standard deviation) scored as the minimal clinically significant difference.
Patient Reported Outcomes - Physical Activity | Up to 6-weeks post-operatively
  Outcome #6 will measure patient reported outcomes and functional status via completion of the computer-adaptive NIH PROMIS measure for physical activity.
  For each of the PROMIS measures, a score of 50 is the average for the United States general population with a standard deviation of 10. All scores are converted to T-scores. The T-score and standard error are automatically reported after completion of the computer-adaptive test. A higher PROMIS T-score represents more of the concept being measured. As each patient will have a pre-operative baseline score, the difference between pre- and post-operative scores will be utilized for all further analysis, with a difference of 10 points (1-standard deviation) scored as the minimal clinically significant difference.
Patient Reported Outcomes - Strength Impact | Up to 6-weeks post-operatively
  Outcome #7 will measure patient reported outcomes and functional status via completion of the computer-adaptive NIH PROMIS measure for strength impact.
  For each of the PROMIS measures, a score of 50 is the average for the United States general population with a standard deviation of 10. All scores are converted to T-scores. The T-score and standard error are automatically reported after completion of the computer-adaptive test. A higher PROMIS T-score represents more of the concept being measured. As each patient will have a pre-operative baseline score, the difference between pre- and post-operative scores will be utilized for all further analysis, with a difference of 10 points (1-standard deviation) scored as the minimal clinically significant difference.

OTHER OUTCOMES:
Pain-Related Disability and Post-Operative Functional Status. | Up to 6-weeks post-operatively
  Outcome #8 will measure post-operative functional status via a 5-question survey on the following activities: sleeping through the night without awaking for pain medication, walking outside the house, showering and dressing independently, patient return to school and parent return to work. Each of these questions was selected as a proxy for improved functional status. Each question is answered 'Yes' or 'No", and graded '1' or '0', respectively. A higher score represents improved functional status. Each of these questionnaires will be administered on a weekly basis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Diab, MD, Principal Investigator — UCSF Department of Orthopaedic Surgery
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charette S, Fiola JL, Charest MC, Villeneuve E, Theroux J, Joncas J, Parent S, Le May S. Guided Imagery for Adolescent Post-spinal Fusion Pain Management: A Pilot Study. Pain Manag Nurs. 2015 Jun;16(3):211-20. doi: 10.1016/j.pmn.2014.06.004. Epub 2014 Nov 6. PMID 25439116
- [Background] LaMontagne L, Hepworth JT, Salisbury MH, Cohen F. Effects of coping instruction in reducing young adolescents' pain after major spinal surgery. Orthop Nurs. 2003 Nov-Dec;22(6):398-403. doi: 10.1097/00006416-200311000-00005. PMID 14705469
- [Background] Rabbitts JA, Aaron RV, Fisher E, Lang EA, Bridgwater C, Tai GG, Palermo TM. Long-Term Pain and Recovery After Major Pediatric Surgery: A Qualitative Study With Teens, Parents, and Perioperative Care Providers. J Pain. 2017 Jul;18(7):778-786. doi: 10.1016/j.jpain.2017.02.423. Epub 2017 Feb 21. PMID 28232147
- [Background] Rhodes L, Nash C, Moisan A, Scott DC, Barkoh K, Warner WC Jr, Sawyer JR, Kelly DM. Does preoperative orientation and education alleviate anxiety in posterior spinal fusion patients? A prospective, randomized study. J Pediatr Orthop. 2015 Apr-May;35(3):276-9. doi: 10.1097/BPO.0000000000000260. PMID 25036417
- [Background] Connelly M, Fulmer RD, Prohaska J, Anson L, Dryer L, Thomas V, Ariagno JE, Price N, Schwend R. Predictors of postoperative pain trajectories in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2014 Feb 1;39(3):E174-81. doi: 10.1097/BRS.0000000000000099. PMID 24173016